CLINICAL TRIAL: NCT01709968
Title: Magnesium Oxide Monohydrate for Nocturnal Leg Cramps (MgNLC); a Prospective, Randomized, Double Blind, Placebo Controlled Clinical Trial.
Brief Title: Magnesium Oxide Monohydrate for Nocturnal Leg Cramps
Acronym: MgNLC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Blinded interim analysis Recommendation, submitted April 1, 2014, was early termination for futility.
Sponsor: Uzi Milman (Other)
Responsible Party: Sponsor-Investigator, Uzi Milman, Director, Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Com120009ctil
Record Dates: First submitted 2012-10-17; First posted 2012-10-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Nocturnal Leg Cramps; Quality of Life
Keywords: Nocturnal Leg Cramps; Quality of life; Quality of sleep
MeSH Terms: conditions — Sleep-Wake Transition Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAGNOX 520® (Experimental): MAGNOX 520® (un-organic granular magnesium complex, composed of Magnesium Oxide & Magnesium Oxide Monohydrate 865mg, Provides 520 mg of free elemental Mg ++); Oral administration once daily for 4 weeks.
  Interventions: Drug: MAGNOX 520®
- Similarly looking placebo. (Placebo Comparator): Similarly looking placebo. Oral administration once daily for 4 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MAGNOX 520® — un-organic granular magnesium complex, composed of Magnesium Oxide & Magnesium Oxide Monohydrate 865mg, Provides 520 mg of free elemental Mg ++); Oral administration once daily for 4 weeks
  Arms: MAGNOX 520®
Drug: placebo — Similarly looking placebo. Oral administration once daily for 4 weeks
  Other Names: Similarly looking placebo
  Arms: Similarly looking placebo.

SUMMARY:
Nocturnal leg cramps (NLC) are painful, involuntary contractions of muscles occurring at rest, mostly at night. A Cochrane review on leg cramps in pregnancy showed some potential benefits in trials of magnesium. This is a single center, prospective, randomized, double blind, placebo controlled clinical trial that aims to investigate the effect of treatment with Magnox 520® (un-organic granular magnesium complex, composed of Magnesium Oxide & Magnesium Oxide Monohydrate 865mg, Provides 520 mg of free elemental Mg++) on frequency and severity of NLC, quality of sleep and quality of life. Hypothesis: Magnox 520® may reduce the number and severity of NLC; an improvement in the quality of life and quality of sleep may ensue.

DETAILED DESCRIPTION:
Ads in the local media and pharmacies will invite individuals afflicted by NLC to participate in the study. Each participating individual will undergo two weeks of eligibility screening followed by 4-week double-blind treatment. The number, severity and duration of NLC will be measured daily as documented in a designated, structured sleep dairy. Quality of life and quality of sleep will be assessed by SF-36 and PSQI questionnaires, respectively, to be completed twice - at enrollment and within one week of the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent before any procedure or assessment is done. Age over 21 years old. Over 4 episodes of documented NLC during 2 weeks of eligibility screening (for the treatment phase).

Insured by Clalit Health Services (CHS). Hebrew speaking

Exclusion Criteria:

Pregnancy Currently taking Quinidine or Magnesium additive Renal failure - serum creatinine more than 2 mg/DL or estimated glomerular filtration rate (eGFR) less than 60 ml/min (the worst, ascertained by the participant electronic records in the last 6 months). If the result is near these limits (i.e. serum creatinin 1.5-2) a second analysis will be done near the study enrollment.

Major neurological disease- ALS, MS, Paraplegia or Quadriplegia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of documented episodes of NLC | 4 weeks
  The primary efficacy endpoint is the difference in the number of episodes of NLC documented in the NCSD, as compared between the MAGNOX 520® and the placebo treated individuals, during a treatment period of 4 weeks;

SECONDARY OUTCOMES:
Severity of documented episodes of NLC | 4 weeks
  The difference in the severity of episodes of NLC documented in the NCSD, as compared between the MAGNOX 520® and the placebo treated individuals, during a treatment period of 4 weeks;
Duration of documented episodes of NLC documented | 4 weeks
  The difference in the duration of episodes of NLC documented in the NCSD, as compared between the MAGNOX 520® and the placebo treated individuals, during a
Quality of life | 4 weeks
  The difference in the change in quality of life (measured by SF36 at enrolment and after the treatment period) between the MAGNOX 520® and the placebo treated individuals;
Quality of sleep | 4 weeks
  The difference in the change in quality of sleep (measured by PSQI at enrolment and after the treatment period) between the MAGNOX 520® and the placebo treated individuals;

CONTACTS AND LOCATIONS:
Overall Officials: Noga Maor Rougin, MD, Principal Investigator — Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District, HAIFA, ISRAEL; Uzi Milman, MD, Study Director — Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District, HAIFA, ISRAEL
Locations (1):
- Clinical Research Unit, Clalit Health Services, Haifa and Western Galilee District,, Haifa, Israel

REFERENCES:
- [Result] Roguin Maor N, Alperin M, Shturman E, Khairaldeen H, Friedman M, Karkabi K, Milman U. Effect of Magnesium Oxide Supplementation on Nocturnal Leg Cramps: A Randomized Clinical Trial. JAMA Intern Med. 2017 May 1;177(5):617-623. doi: 10.1001/jamainternmed.2016.9261. PMID 28241153
- [Derived] Luo L, Zhou K, Zhang J, Xu L, Yin W. Interventions for leg cramps in pregnancy. Cochrane Database Syst Rev. 2020 Dec 4;12(12):CD010655. doi: 10.1002/14651858.CD010655.pub3. PMID 33275278
- See also: pubmed/28241153 — https://www.ncbi.nlm.nih.gov/pubmed/28241153